CLINICAL TRIAL: NCT04576572
Title: Comparison of Criteria for Liver Transplantation in Hepatocellular Carcinoma
Status: Completed | Type: Observational
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Volkan Ince, Assoc.Prof., Inonu University
Other Study IDs: LT-Criteria-HCC
Record Dates: First submitted 2020-09-30; First posted 2020-10-06 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-09

CONDITIONS: Hepatocellular Carcinoma; Liver Cancer; Advanced Adult Hepatocellular Carcinoma; Cirrhosis, Liver; Unresectable Liver Cancer; Liver Transplant Disorder
Keywords: Hepatic malignancy; malignancy; living donor; liver transplantation; expanded criteria; extended; liver cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms; Liver Cirrhosis; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hepatocellular cancer is the 6th most common seen disease in the world and the 3rd in cancer-related deaths. Liver transplantation is the primary curative treatment of HCC, as it eliminates liver cancer and underlying cirrhosis. However, liver transplantation is not offered to every HCC patient, since advanced stage HCC patients are lost with tumor recurrence early after liver transplantation. The Milan criteria, which are accepted worldwide, are the patient selection criteria that we have to follow in cadaver-to-liver transplantation for HCC in our country. However, as the Milan criteria are very strict criteria, it pushes patients out of liver transplantation who exceed the Milan criteria but who can benefit from liver transplantation. Liver transplantation centers all over the world have declared their own criteria under the expanded Milan criteria. In our country, Malatya Criteria have been defined by İnönü University on this subject, and our studies on this subject still continue. When we scan the original articles of all these defined criteria, incomplete data are formed and therefore the strength of the criteria cannot be clearly revealed. For this reason, we aimed to analyze the results of our center and present information about the power of the criteria to the literature.

DETAILED DESCRIPTION:
Aim: To investigate the criteria with the longest overall and disease-free survival and lowest recurrence rates in liver transplantation for hepatocellular cancer (HCC).

Introduction: When the liver transplant criteria for HCC were examined, we saw that many criteria defined in their original articles did not include the rates of extending the Milan criteria, survival and recurrence rates of non-milan patients who were within the newly defined criteria. Therefore, information on which of the criteria defined for liver transplantation in HCC extends the Milan criteria more, which has a longer survival rate and which has a lower recurrence rate is lacking. In order to eliminate this deficiency or at least to have a rough idea, we aimed to compare the results of liver transplantation, performed for HCC in our institute which is a high-volume liver transplant center, by analyzing it according to the existing defined criteria. Thus, we were able to compare the criteria in a homogeneous patient group that was formed as a result of the same inclusion and exclusion criteria in the same period of time. The highest overall and disease-free survival, the lowest recurrence rate, and the criterion that extends the Milan criteria will be introduced. In addition, this study is the first comprehensive comparison of liver transplant criteria for HCC.

Methods: Between March 2002 and July 2020, the data of 424 patients who underwent liver transplantation due to HCC at the Liver Transplantation Institute of İnönü University will be retrospectively analyzed from the prospectively recorded data bank and automation system. Tumor size, tumor number, differentiation and microscopic venous invasion data will all be recorded from the data in the explant pathology report. Since the primary aim of our study is cancer-related survival in patients who can be transplanted, 31 patients with tumor invasion outside the liver (extrahepatic portal vein tumor thrombosis, perihilar lymph node metastasis, diaphragmatic invasion etx) and 70 patients with follow-up period after liver transplantation below 90 days will be excluded from the study. The remaining 323 patients will be included in the study and their data will be analyzed. First, demographic data, tumor characteristics, overall and disease-free survival and recurrence rate of 323 HCC patients who were the study group, will be calculated, and then these patients will be divide groups according to be within or beyond the criteria, than survival and recurrence rates will be calculated. It was then examined whether these expanded criteria actually extended the Milan criteria. It was checked whether a defined Expanded criterion allowed liver transplantation for patients outside of Milan while excluding patients within Milan from liver transplantation. How far the expanded criteria expand the Milan and survival of the patients who beyond Milan but within the criteria were analyzed separately. Thus, the most useful criterion for liver transplantation in HCC treatment will be revealed.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergone liver transplantation due to hepatocellular carcinoma
* Incidentally detected hepatocellular carcinoma at the explant pathology report

Exclusion Criteria:

* Patients with follow up period below 90 days
* Advanced Tumors which have lymph node positivity, main PV tumor thrombosis, adjacent tissue invasion defined by explant pathology etc.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Between 2002 - 2020 August, patients undergone Liver Transplantation at Liver Transplant Institute of Inonu University.
Sampling Method: Non-Probability Sample
Enrollment: 424 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Disease Free Survival | five years
  Tumor free survival after liver transplantation
Overall Survival | five years
  Overall survival after liver transplantation
Tumor recurrence | 5 year
  Tumor recurrence following liver transplantation

SECONDARY OUTCOMES:
The Best Criteria | 5 years
  Liver Transplant criteria which has the best survivals

CONTACTS AND LOCATIONS:
Overall Officials: Volkan Ince, MD, Principal Investigator — Inonu University, Liver Transplant Institute
Locations (1):
- Liver Transplantation Institute, Inonu University, Malatya, Battalgazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in publication
Supporting Information: Study Protocol, SAP
Time Frame: 01.01.2022